CLINICAL TRIAL: NCT06244628
Title: Safety and Efficacy of Iguratimod in the Treatment of Chronic GVHD After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Safety and Efficacy of Iguratimod in the Treatment of Chronic GVHD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, professor, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2023-KL371-01
Record Dates: First submitted 2024-01-26; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: cGVHD
Keywords: Iguratimod; cGVHD
MeSH Terms: interventions — iguratimod

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iguratimod (Experimental): Oral administration of Iguratimod, 25mg twice daily.
  Interventions: Drug: Iguratimod

INTERVENTIONS:
Drug: Iguratimod — Oral administration of Iguratimod, 25mg twice daily

SUMMARY:
This is a randomized, single-center phase 3 clinical trial without blinding. Iguratimod, as a rheumatoid arthritis medication, is used to treat autoimmune diseases such as Sjögren's syndrome. It has acceptable side effects, good clinical availability, and is cost-effective. The investigators plan to recruit participants for a clinical trial to evaluate the efficacy and safety of Iguratimod in the treatment of chronic GVHD.

DETAILED DESCRIPTION:
The investigators plan to recruit participants for a clinical trial to evaluate the efficacy and safety of Iguratimod in the treatment of chronic GVHD. Iguratimod possesses anti-inflammatory, anti-bone resorption, immune modulation, and anti-fibrotic effects. Considering that the pathogenesis of chronic GVHD involves inflammation, immune dysregulation, and fibrosis, Iguratimod is theoretically a potential treatment for cGVHD. In animal experiments, Iguratimod has demonstrated the ability to alleviate glandular inflammation, inhibit BAFF activity, reduce antibody production, and mitigate lung fibrosis. These findings provide a basis for Iguratimod's potential use in the treatment of cGVHD based on animal experimentation. In clinical practice, Iguratimod has been shown to alleviate dry mouth and dry eye symptoms in patients with Sjögren's syndrome. Since cGVHD shares similar symptoms of dry mouth and dry eye, with mechanisms resembling those in Sjögren's syndrome, it is reasonable to infer that Iguratimod used in the treatment of cGVHD patients could alleviate these symptoms and improve their quality of life. Similarly, organ damage in the lungs of cGVHD patients is mainly manifested as TGF-β activation-induced interstitial changes and pulmonary fibrosis. Studies suggest that adding Iguratimod to the treatment of patients with Sjögren's syndrome-induced lung interstitial changes and pulmonary fibrosis can inhibit TGF-β expression, thereby improving lung function and reducing the progression of pulmonary fibrosis. Therefore, the investigators hypothesize that Iguratimod is also effective against cGVHD-induced pulmonary fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years who have undergone allogeneic hematopoietic stem cell transplantation (allo-HSCT), regardless of gender.
2. Those with persistent manifestations of chronic graft-versus-host disease (cGVHD) and suitable for systemic treatment.
3. Previously received at least 1 but not more than 5 lines of systemic treatment for cGVHD.
4. Corticosteroid therapy dose stable for the two weeks before screening; or, if taking prednisone or an equivalent dose of other corticosteroids at a dose >0.5mg/kg/day for four weeks, with ongoing cGVHD manifestations and no improvement; or, if two attempts to taper steroids to a lower dose have failed, and it is necessary to increase the prednisone dose to >0.25mg/kg/day or an equivalent dose.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score: 0~1.
6. Anticipated survival of more than 12 months.

   General criteria:
7. Serum pregnancy test negative for women of childbearing age during the screening period.
8. Sexually active women of childbearing age participating in this study must agree to contraception during the trial and after the last dose of medication.

Exclusion Criteria:

1. Patients who have received experimental treatment for systemic cGVHD within the 28 days prior to enrollment, which was effective and could completely alleviate immunosuppression.
2. Blood cancer relapse (according to the corresponding criteria for relapse of the primary blood cancer) or post-transplant lymphoproliferative disease at the time of screening.

   Laboratory tests:
3. Absolute neutrophil count (ANC) <1.5×10^9/L (excluding GVHD as the cause).
4. Platelet count <50×10^9/L (excluding GVHD as the cause).
5. Alanine aminotransferase (ALT) >3 times the upper limit of normal (ULN), aspartate aminotransferase (AST) >3×ULN (excluding GVHD as the cause).
6. Total bilirubin (TBIL) >1.5×ULN (excluding GVHD as the cause).
7. Creatinine clearance CrCl <60 mL/min (Cockcroft-Gault formula).

   General criteria:
8. Pregnant or lactating women.
9. History of serious illness or other evidence indicating a serious illness, or any other condition that the investigator believes may make the subject unsuitable for this study.

   * History of severe cardiovascular disease [New York Heart Association (NYHA) functional class III or IV], including but not limited to ventricular arrhythmias requiring clinical intervention, uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg); within 6 months prior to enrollment, there is unstable angina, acute coronary syndrome, congestive heart failure, stroke, or other cardiovascular events of class III or above; at screening, NYHA functional class ≥II or left ventricular ejection fraction (LVEF) <50% on echocardiography.
   * Unable to take oral medications, with severe (NCI CTCAE v5.0 ≥ grade 3) chronic gastrointestinal dysfunction, the presence of malabsorption syndrome, or any other condition affecting gastrointestinal absorption.
   * History of clear neurological or psychiatric disorders (including epilepsy or dementia), currently suffering from psychiatric disorders, or judged by the investigator to be non-compliant and unsuitable for participation in the study.
   * History of other severe (NCI CTCAE v5.0 ≥ grade 3) systemic diseases, deemed unsuitable for participation in the clinical trial by the investigator.
10. Other circumstances in which the investigator deems it inappropriate to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Baseline up to 60 days after taking Iguratimod
  Adverse events assessed according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
complete response (CR) | Month 1, 2, 3 and 4
  Assessment of CR at Month 1, 2, 3 and 4. According to the CHRONIC GVHD ACTIVITY ASSESSMENT - CLINICIAN recorded in NIH Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. The 2014 Response Criteria Working Group report. (Biol Blood Marrow Transplant. 2015 Jun;21(6):984-99.)
partial response (PR) | Month 1, 2, 3 and 4
  Assessment of CR at Month 1, 2, 3 and 4. According to the CHRONIC GVHD ACTIVITY ASSESSMENT - CLINICIAN recorded in NIH Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. The 2014 Response Criteria Working Group report. (Biol Blood Marrow Transplant. 2015 Jun;21(6):984-99.)
stable disease (SD) | Month 1, 2, 3 and 4
  Assessment of SD at Month 1, 2, 3 and 4. According to the CHRONIC GVHD ACTIVITY ASSESSMENT - CLINICIAN recorded in NIH Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. The 2014 Response Criteria Working Group report. (Biol Blood Marrow Transplant. 2015 Jun;21(6):984-99.)
progressed disease (PD) | Month 1, 2, 3 and 4
  Assessment of PD at Month 1, 2, 3 and 4. According to the CHRONIC GVHD ACTIVITY ASSESSMENT - CLINICIAN recorded in NIH Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. The 2014 Response Criteria Working Group report. (Biol Blood Marrow Transplant. 2015 Jun;21(6):984-99.)

CONTACTS AND LOCATIONS:
Locations (1):
- Kailin Xu, Xuzhou, Jiangsu, China